CLINICAL TRIAL: NCT02506946
Title: Nonalcoholic Fatty Liver Disease (NAFLD), Insulin Resistance and Dyslipidemia in Adolescents and Young Adults With Polycystic Ovary Syndrome (PCOS)
Brief Title: NAFLD in Adolescents and Young Adults With PCOS
Status: Suspended | Type: Observational
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAA7793
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Polycystic Ovary Syndrome; Non-Alcoholic Fatty Liver Disease; Metabolic Syndrome
Keywords: Polycystic Ovary Syndrome; Non-Alcoholic Fatty Liver Disease; Adolescents; Young Women; MRI; MRS; DXA; Hirsutism; Amenorrhea; Metabolic syndrome; Dyslipidemia; Percentage liver fat
MeSH Terms: conditions — Polycystic Ovary Syndrome; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Hirsutism; Amenorrhea; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples will be stored in a freezer for assays requiring batch testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS subjects: Forty adolescents and young adults between the ages of 14 and 25 years with Polycystic Ovary Syndrome (PCOS) at least two years past menarche.
- Control subjects: Forty unaffected adolescents and young adults between the ages of 14 and 25 years at least two years past menarche.

SUMMARY:
This project focuses on an at-risk adolescent and young adult population who may gain long-term health benefits from detection of risk factors at a young age. The primary aims of this proposal are: 1) To observe whether adolescents and young adults with Polycystic Ovary Syndrome (PCOS) are more likely to have elevated liver fat (>/=4.8%) than controls by studying liver fat deposition measured by magnetic resonance spectroscopy (MRS); 2) To assess the association of percentage liver fat with biomarkers of Non-alcoholic fatty liver disease (NAFLD), dyslipidemia, insulin resistance and body composition in PCOS and controls.

In the proposed study, 40 adolescents and young adults with PCOS and 40 age-comparable control subjects will be evaluated for metabolic disturbances and elevated liver fat using noninvasive and state-of-the-art techniques including MRI, dual-energy x-ray absorptiometry and an oral glucose tolerance test in order to fully assess the metabolic and body composition differences between these groups. This research proposal represents a critical step in understanding the metabolic and cardiovascular comorbidities of PCOS and their relationship to NAFLD. The investigator hopes to use the results generated by this research proposal in order to lay the groundwork for the prevention and treatment of metabolic disorders in adolescents with PCOS. The overarching goal is to decrease and prevent lifelong morbidity associated with this common disorder.

DETAILED DESCRIPTION:
PCOS is a common condition that frequently presents in adolescence and young adulthood and is defined by the presence of hyperandrogenism and ovulatory dysfunction. Affected individuals are at increased risk of insulin resistance, NAFLD and dyslipidemia, which are features associated with the metabolic syndrome, a major public health concern. The associations between PCOS and both insulin resistance and dyslipidemia have been extensively described; however, its association with NAFLD has only recently been noted and superficially studied in adolescents and young adults. Additionally, it has not yet been fully elucidated why seemingly healthy nonobese adolescents with PCOS are predisposed to insulin resistance and its related complications. The susceptibility of certain PCOS patients to developing NAFLD is theorized to be due to the following potentiating factors: insulin resistance, hyperandrogenemia, and a genetic predisposition.

ELIGIBILITY:
Inclusion Criteria:

* All: Healthy; between 14 and 25 years; at least 2 years postmenarche
* PCOS: Clinical hyperandrogenism and/or hyperandrogenemia, menstrual dysfunction (oligomenorrhea or amenorrhea) and exclusion of other known disorders. PCOS will be diagnosed using the NIH 1990 criteria.
* Controls: Regular menses; no clinical hyperandrogenism and/or hyperandrogenemia

Exclusion Criteria:

* Past or present history of a medical disorder or medication known to affect body composition, insulin secretion and sensitivity, or the growth hormone (GH)-insulin-like growth factor 1 (IGF1) axis (eg steroid hormone or thyroid replacement).
* History of current or past pregnancy
* Hormonal contraceptive or metformin use within 3 months of enrollment
* Nonclassical congenital adrenal hyperplasia

Ages: 14 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy adolescent girls and young women 14 - 25 years with and without PCOS
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-07; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Difference in percentage liver fat between PCOS and controls in adolescents and young adults | 1 day
  To compare percentage liver fat by magnetic resonance spectroscopy between adolescents and young adults with PCOS and controls to determine if there is a difference between these groups.

SECONDARY OUTCOMES:
The association of percentage liver fat by magnetic resonance spectroscopy with insulin resistance as measured by HOMA-IR. | 1 day
  The association of percent liver fat with insulin resistance as measured by HOMA-IR will be measured by correlation/regression.
The association of percentage liver fat by magnetic resonance spectroscopy with triglycerides | 1 day
  The association of percent liver fat with triglycerides will be measured by correlation/regression.
The association of percentage liver fat by magnetic resonance spectroscopy with visceral adipose tissue (VAT) | 1 day
  The association of percent liver fat with visceral adipose tissue (VAT) will be measured by correlation/regression.
The association of percentage liver fat by magnetic resonance spectroscopy with total body adipose tissue | 1 day
  The association of percent liver fat with total body adipose tissue will be measured by correlation/regression.

CONTACTS AND LOCATIONS:
Overall Officials: Aviva Sopher, MD, MS, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will consider this

REFERENCES:
- [Background] Sopher AB, Grigoriev G, Laura D, Cameo T, Lerner JP, Chang RJ, McMahon DJ, Oberfield SE. Anti-Mullerian hormone may be a useful adjunct in the diagnosis of polycystic ovary syndrome in nonobese adolescents. J Pediatr Endocrinol Metab. 2014 Nov;27(11-12):1175-9. doi: 10.1515/jpem-2014-0128. PMID 25003376
- [Background] Sopher AB, Gerken AT, Blaner WS, Root JM, McMahon DJ, Oberfield SE. Metabolic manifestations of polycystic ovary syndrome in nonobese adolescents: retinol-binding protein 4 and ectopic fat deposition. Fertil Steril. 2012 Apr;97(4):1009-15. doi: 10.1016/j.fertnstert.2012.01.111. Epub 2012 Feb 17. PMID 22341881
- See also: Information about PCOS — http://womenshealth.gov/publications/our-publications/fact-sheet/polycystic-ovary-syndrome.html
- See also: Information about NAFLD — http://www.liverfoundation.org/abouttheliver/info/nafld/